CLINICAL TRIAL: NCT00002308
Title: A Randomized Blinded Evaluation of Two Doses of Stavudine (2',3'-Didehydro-2',3'-Dideoxythymidine; d4T) to Make Treatment Available to Severely Immunocompromised Patients With HIV Infection Who Have Failed or Are Intolerant of Alternative Antiretroviral Therapy
Brief Title: A Study of Stavudine in HIV-Infected Patients Who Have Not Had Success With Other Anti-HIV Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 116B; AI455-900
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Stavudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Stavudine

INTERVENTIONS:
Drug: Stavudine

SUMMARY:
To make stavudine (d4T) available to patients with advanced HIV disease for whom no alternative antiretroviral is satisfactory. To study the safety and efficacy of two dose levels in a twice-daily regimen.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV positivity with CD4 count < 300 cells/mm3.
* Intolerance to or failure on approved antiretroviral therapy.
* Ability to provide informed consent (of parent or guardian if appropriate).

NOTE:

* Incarcerated persons may be eligible to participate.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Grade 2 or worse disease-related peripheral neuropathy.
* Unresolved drug-related peripheral neuropathy of any severity that is attributable to other nucleoside analogs (AZT, ddC, ddI).
* Malignancy likely to require systemic chemotherapy with myelosuppressive or neurotoxic drugs in the first 3 months of stavudine treatment.
* Pregnancy (physicians of pregnant patients may contact Bristol-Myers to determine eligibility for stavudine therapy in another protocol).

Strongly discouraged:

* AZT, ddI, ddC, and other antiretroviral agents.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 1991-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol - Myers Squibb Co, Princeton, New Jersey, United States